CLINICAL TRIAL: NCT06556992
Title: Fitness Integrative Training for Pediatric Rheumatology Disorders (FIT Teens II): a Pilot Feasibility Study
Brief Title: Fitness Integrative Training for Pediatric Rheumatology Disorders
Acronym: FIT Teens 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIN002FIT-Teens2
Record Dates: First submitted 2024-08-09; First posted 2024-08-16 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Juvenile Idiopathic Arthritis; Systemic Lupus Erythematosus of Childhood; Joint Hypermobility; Juvenile Dermatomyositis
MeSH Terms: conditions — Arthritis, Juvenile; Joint Instability; Dermatomyositis

STUDY DESIGN:
Intervention Model Description: Single arm behavioral intervention feasibility trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FIT Teens (Experimental): Fitness Integrative Training for Teens (FIT Teens) is a combined coping skills training and physical exercise program. Pain coping skills training, also called cognitive behavioral therapy (CBT) teaches a number of behavioral skills (e.g. breathing, relaxation, activity pacing, distraction, and calming statements). Participants also receive a specialized type of neuromuscular exercise training which focuses on core strength, gait and balance.
  Interventions: Behavioral: FIT Teens

INTERVENTIONS:
Behavioral: FIT Teens — This intervention will consist of 16 in-person and remote group-based sessions held twice per week over 8 weeks. Sessions last 90 minutes and will be led jointly by a psychologist/therapist and exercise trainer using manualized protocols.

SUMMARY:
This study evaluates the feasibility of the Fitness Integrative Training program for Teens (FIT Teens 2), a combined cognitive behavioral therapy and neuromuscular exercise training program in patients with pediatric rheumatic diseases and/or joint hypermobility.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric rheumatic diseases (PRD) or joint hypermobility (JH) diagnosed by a pediatric rheumatologist or pain physician.
* Initial diagnosis ≥ 3 months ago
* Ages 10-19 years, inclusive
* Ongoing symptoms of musculoskeletal pain and/or fatigue for at least 3 months
* Functional Disability Index (FDI) Score ≥ 13 indicating at least moderate disability.
* Child has written and spoken proficiency in English and parent has written and spoken proficiency in English or Spanish (will have a certified bilingual provider or interpreter available)

Exclusion Criteria:

* Untreated major psychiatric diagnoses (e.g., major depression, bipolar disorder, psychoses) or documented developmental delay.
* Any other medical condition determined by their physician to be a contraindication for exercise.
* Childhood Myositis Assessment Scale (CMAS) ≤ 30

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2024-09-24 (Actual); Primary Completion 2025-07-02 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of Enrollment | 2 years
  Maintain consistent monthly enrollment for the duration of the project
Session Attendance | 8 weeks
  Evaluation of the number of sessions attended out of the 16 sessions offered
Participant Retention at Post-Treatment | 8 weeks
  Number of participants completing post-treatment visit
Treatment Fidelity | 2 years
  All sessions will be video-recorded and trainers adherence to the protocol will be assessed using an 9-item fidelity checklist (e.g., homework and diary review, CBT skill instruction and practice, neuromuscular exercise instruction and practice, CBT and exercise homework planning).
Participant Safety | 2 years
  Assessment of frequency and severity of adverse events possibly, likely, or definitely related to the study treatment or procedures

CONTACTS AND LOCATIONS:
Overall Officials: Susmita Kashikar-Zuck, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States